CLINICAL TRIAL: NCT02305810
Title: An Angiogenic Study in Patients With Well/Moderately Differentiated Metastatic Pancreatic Neuroendocrine Tumors Treated With Everolimus
Brief Title: A Biological Prospective Study in Patients With Metastatic Pancreatic NETs Treated With Everolimus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: S543/310
Record Dates: First submitted 2014-06-17; First posted 2014-12-03 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-09

CONDITIONS: Pancreatic Neuroendocrine Tumour Metastatic
MeSH Terms: interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm receiving everolimus (Experimental): single treatment arm receiving everolimus 10 mg daily
  Interventions: Drug: Everolimus 10 mg daily

INTERVENTIONS:
Drug: Everolimus 10 mg daily — everolimus is a recently approved mTOR inhibitor in advanced progressing well/moderately differentiated pancreatic neuroendocrine tumors
  Other Names: RAD 001

SUMMARY:
Everolimus represents an approved therapy for patients with advanced well/moderately differentiated pancreatic NETs. Although some patients could benefit from this drug in terms of long-term tumor growth control, others are resistant upfront or become resistant during treatment. Therefore, it is crucial to detect some biological factors which can help to identify the responsive tumors. Given that Everolimus is a biological agent and its mechanism of action can be partially directed towards angiogenesis its effects can be studied on different levels and with different methods. Upfront and early surrogate predictive markers of activity/efficacy can be studied on tumor tissue, tumor imaging, and peripheral blood. mTOR pathways alterations, circulating endothelial cells, and other circulating angoigenic factors will be correlated with clinical outcome. Tumor perfusion and circulating markers will be studied also as markers of response compared with the morphological imaging.

DETAILED DESCRIPTION:
• Background:: Everolimus has been reported to be effective compared with placebo in well/moderately differentiated pancreatic NETs in terms of progression-free survival (PFS) improvement. However, a number of patients are refractory upfront or become resistant after few months of therapy. Therefore, it is crucial to detect some biological factors which can help to identify the responsive tumors. Everolimus is a biological agent and its mechanism of action can be partially directed towards angiogenesis. This can be studied on different levels and with different methods. Upfront and early surrogate predictive markers of activity/efficacy can be studied on tumor tissue, on tumor imaging, and on the peripheral blood. Tumor study with diffusion-MRI and angiogenic circulating markers can be studied also as markers of response compared with the morphological imaging.

* Material and Methods :

  1. Circulating Endothelial Cells (CECs) and Circulating endothelial progenitors (CEPs) will be performed by flow cytometry. The monoclonal antibodies used for the search of CECs and CEPs include: cluster of differentiation antigen 45 (CD45), CD31, CD133, CD146, CD34, VEGFR-2, 7-amino-actinomycin D (7-AAD) and Syto1. Vascular endothelial growth factor (VEGF), basic fibroblast growth factor (bFGF), VEGFR-2 and thrombospondin-1 (TSP-1) will be also detected on the peripheral blood.
  2. On the tumor tissue the following determinations will be performed, including:

     * Subtype 2 somatostatin receptor,
     * Phospho-AKT
     * Phospho-mTOR
     * Phospho-4E-BP1
     * Phospho-p70-S6 kinase Rabbit anti-tuberous sclerosis complex 2 (TSC2) Cell Signaling Technology
     * Mouse anti-PTEN Cell Signaling Technology
  3. Diffusion-weighted imaging (DWI) has been shown to be able to provide information regarding the cellular density and properties of the extracellular matrix and the apparent diffusion coefficient (ADC) value calculated using DWI can serve as a marker of cellularity. Given that tumor cellularity is contributed largely by cellular proliferation, the ADC value can be a surrogate biomarker for tumor-cell proliferation . ADC-Magnetic Resonance Imaging (MRI) will be performed at baseline, after 1 month and after three months of therapy.
* Study design

Baseline, after 1 month of therapy, after three months of therapy and at progression:

* Abdomen DWI-MRI
* CEC, CEPs
* Circulating VEGF, VEGFR-2, bFGF, TSP-1

Baseline biopsy of a metastatic site and possibly a new biopsy at the time of tumor progression

Correlation of biological parameters with clinical outcome ( tumor response and progression free survival, Response Evaluation Criteria in Solid Tumors , RECIST 1.0 criteria)

• Statistical analysis: This is an exploratory study on the potential predictive value of some biological factors (CECs, VEGF and bFGF among them) expressed in terms of reducing risk of progression in patients with advanced pancreatic NETs treated with Everolimus.

We will use two-tailed log-rank test (α = 0.05, 1-β = 0.20) to test the hypothesis of 30% a reduction in risk (hazard rate; HR) equal to HR = 0.30 for those belonging to the following layers:

* ≥ 2.2/uL vs < 2.2/uL for CEC at basal or
* ≤ 65.6 vs > 65.6 for FGF levels after two months since start treatment or
* ≤ 32.5 vs > 32.5 for VEGF levels after two months since start treatment The sample size is calculated to compensate for the power loss of the log-rank test assuming an average and uniform log-rank test drop-out of 10% and bearing in mind that the threshold values refer to the 25th, 75th and 50th percentile distributions of CEC, bFGF, and VEGF, respectively. Considering an accrual rate of 20 patients/year, a treatment period of 12 weeks with a follow-up of 1 year and for a sample size equal to 43 patients, the study will have a total length of about 3 years and 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Histological diagnosis of metastatic well/moderately differentiated pancreatic neuroendocrine tumor
2. Patient incoming to be treated with everolimus outside clinical trials or within a clinical trial that permits the concurrent inclusion in an ancillary trial
3. Written informed consent must be signed and dated by the patient and the investigator prior to inclusion.

Exclusion Criteria:

1. Patients with poorly differentiated neuroendocrine carcinoma, adenocarcinoid, goblet cell carcinoid, small cell carcinoma, Merkel cell carcinoma.
2. Patients with pancreatic NETs not eligible to be treated with everolimus
3. Patients with ongoing everolimus treatment
4. Prior therapy with mTOR inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-09; Primary Completion 2017-01-12 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Circulating angiogenic factors, molecular imaging and tumor tissue factors changes during treatment with RAD001 at baseline, week 4, week 12 and at disease progression. | Baseline, week 4, week 12 up to tumor progression
  Angiogenic factors (circulating endothelial cells, CECs; serum VEGF, bFGF, VEGFR-2, TSP-1) determined by serum samples; tumor tissue mTOR pathway alterations determined by Immunohistochemical staining ; ADC (apparent diffusion coefficient) calculated by Magnetic Resonance Imaging (MRI)

SECONDARY OUTCOMES:
Overall survival (OS) | Baseline to death
  Survival status
RR (response rate) , including SD (stable disease) and PR (partial response) | Baseline to best tumor response or unacceptable toxicity
  Clinical and/or radiological response
TTP, time to progression | Baseline to tumor progression or unacceptable toxicity
  Time from baseline to clionical/radiological signs of disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Fazio, MD,PhD, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy